CLINICAL TRIAL: NCT01501162
Title: Effect of Probiotics on Gut-Liver Axis of Alcoholic Liver Disease
Acronym: EPALD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Suk, doctor, assistant professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPALD
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Results first posted 2015-01-27 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-12

CONDITIONS: Alcoholic Liver Disease
Keywords: hepatitis, alcohol
MeSH Terms: conditions — Liver Diseases, Alcoholic; Hepatitis, Alcoholic | interventions — Hepatitis A Vaccines; Ethanol; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alcohol, hepatitis, Placebo (Placebo Comparator): We explored the therapeutic effects of probiotics in patients with alcoholic hepatitis
  Interventions: Drug: alcohol, hepatitis, Placebo
- hepatitis, alcohol, probiotics (Active Comparator): We explored the therapeutic effects of probiotics in patients with alcoholic hepatitis
  Interventions: Drug: hepatitis, alcohol, probiotics

INTERVENTIONS:
Drug: hepatitis, alcohol, probiotics — 7 days of probiotics (1500 mg/day)
  Other Names: LACTOWELL
  Arms: hepatitis, alcohol, probiotics
Drug: alcohol, hepatitis, Placebo — Placebos of the same shape and size were manufactured at Pharmaceutical Corporation.
  Other Names: Placebo
  Arms: alcohol, hepatitis, Placebo

SUMMARY:
Background/Aims:

The investigators explored the therapeutic effects of probiotics in patients with AH.

Methods:

Between September 2010 and April 2012, the investigators conducted a 7-day, double-controlled, randomized, prospective clinical trial comparing the efficacy of probiotics in improving liver enzymes, LPS, pro-inflammatory cytokines. AH was defined as an aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2 and elevated AST (ALT) level with an alcohol consumption history within 48 hours. Patients were randomized to receive 7 days of probiotics (1500 mg/day) or placebo. The levels of liver enzymes, modified Discriminant Function (mDF), LPS, and pro-inflammatory cytokines were checked at baseline and again after therapy.

DETAILED DESCRIPTION:
Background/Aims: Alcoholic hepatitis (AH) is one of the leading causes of liver diseases. Gut-derived microbial lipopolysaccharide (LPS) has been known as a central role in the pathogenesis of AH. Some animal studies suggested an emerging role of probiotics in restoration of the bowel flora and improving liver enzymes. We explored the therapeutic effects of probiotics in patients with AH.

Methods: Between September 2010 and April 2012, we conducted a 7-day, double-controlled, randomized, prospective clinical trial comparing the efficacy of probiotics in improving liver enzymes, LPS, pro-inflammatory cytokines. AH was defined as an aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2 and elevated AST (ALT) level with an alcohol consumption history within 48 hours. Patients were randomized to receive 7 days of probiotics (1500 mg/day) or placebo. The levels of liver enzymes, modified Discriminant Function (mDF), LPS, and pro-inflammatory cytokines were checked at baseline and again after therapy.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic Hepatitis

Exclusion Criteria:

* Cancer
* Viral Hepatitis, other Hepatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Suk, PhD, Principal Investigator — Department of Internal Medicine, Hallym University Chuncheon Sacred Heart Hospital
Locations (1):
- Department of Internal Medicine, Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, South Korea

REFERENCES:
- [Derived] Han SH, Suk KT, Kim DJ, Kim MY, Baik SK, Kim YD, Cheon GJ, Choi DH, Ham YL, Shin DH, Kim EJ. Effects of probiotics (cultured Lactobacillus subtilis/Streptococcus faecium) in the treatment of alcoholic hepatitis: randomized-controlled multicenter study. Eur J Gastroenterol Hepatol. 2015 Nov;27(11):1300-6. doi: 10.1097/MEG.0000000000000458. PMID 26302024

RESULTS

PARTICIPANT FLOW:
Groups:
- Alcohol, Hepatitis, Placebo: Placebo (for probiotics) for 7 days Placebos of the same shape and size were manufactured at Pharmaceutical Corporation.
Period: Overall Study
Arm/Group | Alcohol, Hepatitis, Placebo | Hepatitis, Alcohol, Probiotics
Started | 65 | 65
Completed | 57 | 60
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol, Hepatitis, Placebo | Hepatitis, Alcohol, Probiotics | Total
Number analyzed (Participants) | 57 | 60 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 60 | 117
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (12.4) | 52.7 (9.4) | 52.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 20 | 22 | 42
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 57 | 60 | 117

OUTCOME MEASURES:

1. Primary Outcome: Liver Enzymes(ALT)
Description: Blood analysis was performed using standard methodologies.
Time Frame: 7 days after probiotics
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Alcohol, Hepatitis, Placebo | Hepatitis, Alcohol, Probiotics
Number analyzed (Participants) | 57 | 60
IU/L | 66 (136) | 48 (49)

2. Secondary Outcome: Lipopolysaccharide (LPS) and Pro-inflammatory Cytokines
Description: For the measurements of cytokines, homogenates of serum were processed with Human Tumor necrosis factor-alpha ELISA Kit and Human interleukin 1 beta ELISA Kit . For the measurement of LPS ELISA Kit was used. Assays were performed according to the manufacturer's instructions.
Time Frame: 7 days after probiotics
Measure: Mean (Standard Deviation); unit: EU/mL
Arm/Group | Alcohol, Hepatitis, Placebo | Hepatitis, Alcohol, Probiotics
Number analyzed (Participants) | 57 | 60
EU/mL | 2.1 (2.7) | 1.7 (1.6)

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed
Arm/Group | Alcohol, Hepatitis, Placebo | Hepatitis, Alcohol, Probiotics
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No